CLINICAL TRIAL: NCT05388123
Title: A Single Arm Phase II Pilot Study of Low Dose Vemurafenib Plus Rituximab in the Front-line and Relapsed/Refractory Treatment of Hairy Cell Leukemia
Brief Title: Low Dose Vemurafenib and Rituximab in Hairy Cell Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-7787
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-12

CONDITIONS: Hairy Cell Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Vemurafenib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low dose Vemurafenib and Rituximab (Experimental): Eligible patients will receive vemurafenib at a dose of 240 mg orally twice daily (b.i.d.) continuously for 8 weeks. Rituximab 375 mg/m2 will be administered every 2 weeks for a total of 16 weeks. The entire duration of treatment will be 16 weeks.
  Interventions: Drug: Low dose vemurafenib plus rituximab

INTERVENTIONS:
Drug: Low dose vemurafenib plus rituximab — Vemurafenib 240 mg twice daily for 8 weeks with concurrent rituximab 375 mg/m2 every 2 weeks followed by maintenance consolidative rituximab 4 times every 2 weeks post-vemurafenib
  Other Names: Vemurafenib; Rituximab

SUMMARY:
The current standard-of-care for Hairy Cell Leukemia involves chemotherapy, with agents such as cladribine or pentostatin. Chemotherapy is associated with infection, low blood counts and predisposition to future cancers. This study tests a new yet previously validated drug combination for the treatment of hairy cell leukemia. The treatment involves 8 weeks of treatment with an oral drug called vemurafenib and 8 doses of an intravenous medication called rituximab. The goal of this study is to see whether this treatment is better tolerated and more effective than the currently used treatment in this disease. In addition, this study uses a lower dose of vemurafenib than previous studies have used, with the goal of minimizing side effects from this medication.

DETAILED DESCRIPTION:
This is a single-center, open label, single arm, investigator-initiated phase II trial of the oral BRAF inhibitor, vemurafenib, plus rituximab in patients with previously untreated or relapsed and refractory HCL. Eligible patients will receive vemurafenib at a dose of 240 mg orally twice daily (b.i.d.) continuously for 8 weeks. Rituximab 375 mg/m2 will be administered concomitantly with vemurafenib every 2 weeks from the first day of treatment. After completion of vemurafenib, the patient will receive rituximab 375 mg/m2 every 2 weeks for a total of 8 weeks. The entire duration of treatment will be 16 weeks. Six months after the initiation of the treatment, a bone marrow aspirate and biopsy will be performed for assessment of response and evaluation of minimal residual disease (MRD).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histologically confirmed HCL that are BRAF V600E positive by IHC or NGS
* Patient's must meet the standard treatment initiation criteria, as defined by ANC ≤1.0, Hgb ≤ 10.0 or PLT ≤100K
* Patients can either have (1) not received any prior therapy for the disease or have had (2) failure to achieve any response to the initial purine analog-based therapy or (3) subsequent relapse after any prior therapy.
* ECOG performance status of 0-2
* Acceptable pre-study organ function during screening not exacerbated by Hairy Cell Leukemia. General thresholds should be a total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN, and serum creatinine ≤ 1.5x ULN
* For women of childbearing potential, agreement to use acceptable methods of contraception
* For men with female partners of childbearing potential, agreement to use barrier contraception
* Negative serum pregnancy test within 7 days of commencement of treatment in premenopausal women.
* Ability to understand and willingness to sign a written informed consent document.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Pregnant or breast-feeding or intending to become pregnant during the study
* Have had chemotherapy (including purine analogs), rituximab, and other investigational agents within six weeks prior to entering the study. The patients cannot have received BRAF inhibitor therapy within 6 months of entering the study.
* Major surgery within 4 weeks prior to entering the study
* Invasive malignancy within the past 2 years prior to first study drug administration, except for adequately treated (with curative intent) basal or squamous cell carcinoma, melanoma, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer or other cancers from which the patient has been disease-free for at least 2 years
* Active HIV, hepatitis B and hepatitis C or any clinically significant history of liver disease. Hepatitis B prior infection is not a contraindication though will require therapy.
* Known hypersensitivity to any of the study drugs
* Patients with HCL that are BRAF V600E mutation negative

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response | Up to 2 years from enrollment
  Resolution of cytopenias and splenomegaly

SECONDARY OUTCOMES:
Time to hematologic response | Up to 2 years from enrollment
  Days until resolution of cytopenias
MRD Status | At 6 months, 1 year and 2 years from treatment
  At the time of bone marrow assessment by testing for BRAFV600E mutation status
Relapse-Free Survival | From start of treatment until 2 years
  Reapperance of Hairy-Cell related cytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Alan Saven, MD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish aggregate data in manuscript

REFERENCES:
- [Background] Tiacci E, De Carolis L, Simonetti E, Capponi M, Ambrosetti A, Lucia E, Antolino A, Pulsoni A, Ferrari S, Zinzani PL, Ascani S, Perriello VM, Rigacci L, Gaidano G, Della Seta R, Frattarelli N, Falcucci P, Foa R, Visani G, Zaja F, Falini B. Vemurafenib plus Rituximab in Refractory or Relapsed Hairy-Cell Leukemia. N Engl J Med. 2021 May 13;384(19):1810-1823. doi: 10.1056/NEJMoa2031298. PMID 33979489
- [Background] Grever M, Andritsos L, Banerji V, Barrientos JC, Bhat S, Blachly JS, Call T, Cross M, Dearden C, Demeter J, Dietrich S, Falini B, Forconi F, Gladstone DE, Gozzetti A, Iyengar S, Johnston JB, Juliusson G, Kraut E, Kreitman RJ, Lauria F, Lozanski G, Parikh SA, Park J, Polliack A, Ravandi F, Robak T, Rogers KA, Saven A, Seymour JF, Tadmor T, Tallman MS, Tam CS, Tiacci E, Troussard X, Zent C, Zenz T, Zinzani PL, Wormann B. Hairy cell leukemia and COVID-19 adaptation of treatment guidelines. Leukemia. 2021 Jul;35(7):1864-1872. doi: 10.1038/s41375-021-01257-7. Epub 2021 May 4. PMID 33947938